# **Statistical Analysis Plan Amendment 4**

**Study ID**: 213171

Official Title of the Study: A phase IIIB, randomized, controlled, observer-blind study to evaluate safety and immunogenicity of GSK's meningococcal ABCWY vaccine when administered in healthy adolescents and adults, previously primed with meningococcal ACWY vaccine.

NCT Number: NCT04707391

**Date of Document:** 15 September 2022

# STATISTICAL ANALYSIS PLAN

# 213171 (MENABCWY-019)

A phase IIIB, randomized, controlled, observer-blind study to evaluate safety and immunogenicity of GSK's meningococcal ABCWY vaccine when administered in healthy adolescents and adults, previously primed with meningococcal ACWY vaccine

**AUTHOR:** PPD

**VERSION NUMBER AND DATE:** 

Final V1.0, 23JUL2020

Final V2.0 (Amendment 1), 14OCT2020

Final V3.0 (Amendment 2), 07APR2021

Final V4.0 (Amendment 3), 10NOV2021

Final V5.0 (Amendment 4), 05SEP2022

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx

Author: PPD Version Number: Final 5.0

# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan Final V5.0 (Dated 05SEP022 for Protocol 213171 (MENABCWY-019), Amendment 3 dated 01NOV2021.

| | Name | Signature | Date (DDMMYYYY) |
|-----------|-----------------------|-----------|-------------------|
| Author: | PPD | PPD<br>R | September 7, 2022 |
| Position: | Statistical Scientist | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMMYYYY) |
|--------------|-----------------------|-------------|-------------------|
| Approved By: | PPD | PPD<br>Ref | September 7, 2022 |
| Position: | Statistical Scientist | · | |
| Company: | IQVIA | | |
| | ' | | |
| Approved By: | PPD | PPD | September 7, 2022 |
| Position: | Expert Statistician | | |
| Company: | GlaxoSmithKline Bio | logicals SA | |
| | ' | | |
| Approved By: | PPD | PPD | September 15, 20 |
| Position: | Lead Statistician | | |
| Company: | GlaxoSmithKline Bio | logicals SA | |

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


# **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| Final 1.0 | 24JUL2020 | 'PPD | Not Applicable – First Version |
| Final 2.0 | 14OCT2020 | | Added APPENDIX 3 for details on protocol deviations and of exclusions from analysis sets |
| Final 3.0 | 05MAR2021 | Updated this document based on the protocol amendment 2 dated 12Feb2021 Changes: Promoted one of the secondary endpoints to coprimary. | |
| Final 4.0 | 10NOV2021 | | Change label of treatment groups in the TFLs Updated this document based on the protocol amendment 3 dated 01NOV2021 Changes: Include potential interim analysis. Include sensitivity analysis Use NHBA strain M13520 |
| Final 5.0 | 05SEP2022 | | Adjust the visit windows for analysis Include information regarding IA process Updated APPENDIX 3 to match latest PDMP Medications coded using WHO-DD rather than GSK DD Update spelling mistakes in APPENDIX 3 |

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Author:

PPD

Final 5.0

05SEP2022

# **TABLE OF CONTENTS**

| 1. | INTR | ODUCTION11 |
|---|---|---|
| 2. | STUD | Y OBJECTIVES AND ENDPOINTS11 |
| 2.1. | Primar | y Immunogenicity Objective11 |
| 2.2. | Second | ary Immunogenicity Objectives11 |
| CCI | | |
| 2.4. | Primar | y Safety Objective |
| 2.5. | Endpoi | nts |
| 2.5 | .1. Pri | mary Immunogenicity Endpoint |
| 2.5 | .2. See | condary Immunogenicity Endpoints |
| CCI | 4 D | |
| 2.5 | .4. Pri | mary Safety Endpoints |
| 3. | STUD | Y DESIGN |
| 3.1. | Genera | l Description16 |
| 3.2. | Schodu | le of Events |
| 3.2. | Schedu | ic of Events10 |
| 3.3. | Change | es to Analysis from Protocol |
| 4. | DI AN | NED ANALYSES19 |
| 4. | FLAN | NED ANALISES19 |
| 4.1. | Data M | onitoring Committee (DMC) |
| | Data M | ontoring commetee (Diric) |
| 4.2. | Interim | Analysis |
| 4.3. | Final A | nalysis19 |
| <b>5.</b> | ANAL | YSIS SETS |
| 5.1. | Process | for Analysis Set Assignment |
| Docur | ment: | C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C |
| | | B4DEE6C228977964.docx |

Version Number:

**CONFIDENTIAL** Version Date:

| 5.2. | Enrolled Set [ENR] |
|---|---|
| 5.3. | Exposed Set [ES] |
| 5.4. | Full Analysis Set [FAS] |
| 5.5. | Per Protocol Analysis Set [PPS] |
| <b>5.6.</b> 5.6. 5.6. 5.6. | 2. Solicited Safety Analysis Set [SSS] |
| 5.7. | Overview of Analysis by Protocol Deviation (PD) |
| 6. | GENERAL CONSIDERATIONS22 |
| 6.1. | Reference Start Date and Study Day |
| 6.2. | Baseline |
| 6.3. | Retests, Unscheduled Visits and Early Termination Data |
| 6.4. | Windowing Conventions |
| 6.5. | Statistical Tests |
| 6.6. | Common Calculations |
| 6.7. | Software Version |
| 7. | STATISTICAL CONSIDERATIONS |
| 7.1. | Adjustments for Covariates and Factors to be Included in Analyses |
| 7.2. | Multicenter Studies |
| 7.3. | Missing data |
| 7.4. | Multiple Comparisons/ Multiplicity |

Document:

Author: Version Number: Final 5.0 PPD

PPD

Author:

| 7.5. | Active-Control Studies Intended to Show Non-inferiority | 27 |
|---|---|---|
| 7.6. | Examination of Subgroups | 27 |
| 7.7. | Randomization and Blinding | 28 |
| 7.7. | | |
| 7.7. | | |
| 8. | OUTPUT PRESENTATIONS | 28 |
| 9. | DISPOSITION AND WITHDRAWALS | 29 |
| 9.1. | Disposition | 29 |
| 9.2. | Protocol Deviations | 29 |
| 10. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 30 |
| 10.1. | Derivations | 30 |
| 11. | VACCINATION AND MEDICAL HISTORY | 31 |
| 12. | CONCOMITANT ILLNESSES | 31 |
| 13. | MEDICATIONS | 32 |
| 14. | STUDY MEDICATION EXPOSURE | 32 |
| 14.1. | Derivations | 32 |
| 15. | STUDY MEDICATION COMPLIANCE | 32 |
| 16. | IMMUNOGENICITY OUTCOMES | 33 |
| 16.1. | Primary Immunogenicity | 33 |
| 16.1 | .1. Primary Immunogenicity Variable & Derivations | 33 |
| 16.1 | | |
| 16.1 | | |
| 16.1 | | |
| 16.1 | .5. Subgroup Analysis of Primary Immunogenicity Variable(s) | 36 |
| 16.2. | Secondary Immunogenicity | 36 |
| Docum | nent: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DIB4DEE6C228977964.docx | DEF7D8D4E7C |

**CONFIDENTIAL** Version Date: 05SEP2022

Final 5.0

Version Number:

| Statistical Analysis Plan | Page 7 of 6 |
|---|---|
| 16.2.1. Secondary Immunogenicity Variables & Derivations | 36 |
| 16.2.1.1. Immune Response, Serogroups A, C, W and Y (measured by hSBA) | |
| 16.2.1.2. Immune Response, Serogroup B Indicator Strains (measured by hSBA) | |
| 16.2.2. Missing Data Methods for Secondary Immonogenicity Variables | |
| 16.2.3. Analysis of Secondary Immunogenicity Variables | |
| 16.2.3.1. Immune Response Analysis, Serogroups A, C, W and Y (measured by hSBA) | 37 |
| 16.2.3.2. Immune Response Analysis, Serogroup B Indicator Strains (measured by hSBA). | |
| 17. SAFETY OUTCOMES | 42 |
| | 12 |
| 17.1. Adverse Events | 42 |
| 17.1.1. Safety Completeness Analysis | |
| 17.1.2. Solicited Events | |
| 17.1.3. Unsolicited Adverse Events | |
| 17.1.4. Combined Solicited and Unsolicited Adverse Events | 48 |
| 17.1.5. COVID-19 Events | 49 |
| 17.2. Laboratory Evaluations | 40 |
| 17.2. Laboratory Evaluations | 49 |
| 18. DATA NOT SUMMARIZED OR PRESENTED | 49 |
| 19. REFERENCES | 50 |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | 51 |
| APPENDIX 2. PARTIAL DATE CONVENTIONS | |
| ADDENDIY 3 DOCTOCOL DEVIATIONS AND EVOLUSIONS EDOM | |

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

ANALYSIS SETS.......58

B4DEE6C228977964.docx


# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ANCOVA | Analysis of covariance |
| ANOVA | Analysis of variance |
| BMI | Body mass index |
| BS | Blood sample |
| CBER | Center for Biologics Evaluation and Research |
| CDER | Center for Drug Evaluation and Research |
| CI | Confidence Interval |
| CSR | Clinical Study Report |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-linked immunosorbent assay |
| ENR | Enrolled Set |
| EoS | End of Study |
| ES | Exposed Set |
| ESFU | Extended safety follow-up |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials Database |
| FAS | Full Analysis Set |
| fHbp | Factor H binding protein |
| GMC | Geometric mean concentration |
| GMR | Geometric mean ratio |
| GMT | Geometric mean titer |
| GSD | Geometric standard deviation |

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


| Abbreviation | Definition |
|---|---|
| GSK | GlaxoSmithKline |
| hSBA | Human Serum Bactericidal Assay |
| ICH | International Council on Harmonisation |
| IgG | Immunoglobulin G |
| LAR | Legally acceptable representative |
| LL | Lower limit |
| LLOQ | Lower limit of quantitation |
| M | Month |
| mm | Millimeter |
| MAR | Missing at random |
| MCAR | Missing completely at random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MenABCWY | Meningococcal serogroups A, B, C, W, and Y investigational vaccine |
| MenACWY | Meningococcal serogroups A, C, W, and Y conjugate vaccine (Menveo) |
| MenB | meningococcal B (Bexsero) |
| NHBA | Neisseria heparin binding antigen |
| NI | Non-inferiority |
| PD | Protocol deviation |
| pIMD | Potential immune-mediated disease |
| PT | Preferred term |
| PPS | Per Protocol Set |
| ROW | Rest of the World |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |

Document:

Author: Version Number: Final 5.0 PPD

# Statistical Analysis Plan


| Abbreviation | Definition |
|--------------|---------------------------|
| SD | Standard deviation |
| SOC | System organ class |
| SSS | Solicited Safety Set |
| Т | Telephone contact |
| USS | Unsolicited Safety Set |
| V | Visit |
| WHO | World Health Organisation |

 $\label{lem:converter} C: \ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7CB4DEE6C228977964.docx$ Document:

Author: Version Number: Final 5.0 PPD

## 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of immunogenicity and safety data for Protocol 213171 (MENABCWY-019). It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol amendment 3.0, dated 01NOV2021.

# 2. STUDY OBJECTIVES AND ENDPOINTS

## 2.1. Primary Immunogenicity Objective

#### Immunological non-inferiority: MenABCWY vs. MenACWY (Family 1):

The first co-primary objective is to demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise (refer to Section 6.6) in human serum bactericidal assay (hSBA) titers against N. *meningitidis* serogroups A, C, W, and Y, at 1 month after the **second** MenABCWY vaccination (0,6-months) and 1 month after the MenACWY vaccination (single dose).

#### Immunological non-inferiority: MenABCWY vs. MenACWY (Family 2):

The second co-primary objective is to demonstrate the immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with a MenACWY vaccine, as measured by the percentages of participants achieving a 4-fold rise (refer to Section 6.6) in hSBA titers against *N. meningitidis* serogroups A, C, W, and Y, at 1 month after the **first** MenABCWY vaccination (0,6-months schedule) and 1 month after the MenACWY vaccination (single dose).

# 2.2. SECONDARY IMMUNOGENICITY OBJECTIVES

The secondary objectives are:

• To assess the immune response to MenABCWY (0,6-month schedule) and MenACWY

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


(single dose) vaccines against *N. meningitidis* serogroups A, C, W, and Y, at pre-vaccination (Day 1, Month 0) and 1 month after the **first and last** MenABCWY vaccinations and 1 month after the MenACWY vaccination.

• To assess the immune response to the MenABCWY vaccine (0,6-month schedule) against *N. meningitidis* serogroup B indicator strains, at pre-vaccination (Day 1, Month 0) at 1 month after the **last** MenABCWY vaccination.

Note: *N. meningitidis* serogroup B indicator strains include: (M14459 for factor H binding protein [fHbp] antigen, M13520 for NHBA antigen, 96217 for NadA antigen and NZ98/254 for PorA P1.4 antigen).



 $\label{loc-converter-app} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


## 2.4. PRIMARY SAFETY OBJECTIVE

The primary safety objective is to evaluate the safety and reactogenicity of the MenABCWY and MenACWY vaccines.

# 2.5. ENDPOINTS

The primary, secondary and tertiary endpoints to support regulatory decisions are described in the following sections.

#### 2.5.1. PRIMARY IMMUNOGENICITY ENDPOINT

#### Immunological non-inferiority: MenABCWY vs. MenACWY (Family 1):

The first co-primary immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine, will be demonstrated if the lower limit (LL) of the 2-sided 95% CI for the group difference in percentages of participants in the PPS (as defined in Section 5.5) achieving a 4-fold rise (refer to Section 6.6) in hSBA titers is above -10%, for each serogroup, i.e., the percentages of participants with a 4-fold rise (refer to Section 6.6) in hSBA titers against N. meningitidis serogroups A, C, W, and Y at 1 month after the **second** vaccination for the ABCWY group (Day 211, Month 7), and 1 month after the single dose of MenACWY vaccination for the ACWY group (Day 31, Month 1), relative to baseline (Day 1, Month 0).

#### Immunological non-inferiority: MenABCWY vs. MenACWY (Family 2):

The second-co-primary immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine, will be demonstrated if the lower limit (LL) of the 2-sided 95% CI for the group difference in percentages of participants in the Per Protocol Analysis Set (PPS, as defined in Section 5.5) achieving a 4-fold rise (refer to Section 6.6) in hSBA titers is above -10%, for each serogroup, i.e., the percentages of participants with a 4-fold rise (refer to Section 6.6) in hSBA titers against *N. meningitidis* serogroups A, C, W, and Y at 1 month after the **first** vaccination for the ABCWY group (Day 31, Month 1), and 1 month after the single dose of MenACWY vaccination for the ACWY group (Day 31, Month 1), relative to baseline (Day 1, Month 0).

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


## 2.5.2. SECONDARY IMMUNOGENICITY ENDPOINTS

The immune response to MenABCWY (0,6-month schedule) and MenACWY (single dose) vaccines against *N. meningitidis* serogroups A, C, W, and Y, at pre-vaccination (Day 1, Month 0) and 1 month after the **first and last** MenABCWY vaccinations and 1 month after the single MenACWY vaccination will be demonstrated for participants in the Full Analysis Set (FAS, as defined in Section 5.4) by:

- The percentages of participants with hSBA titers ≥Lower Limit of Quantitation (LLOQ) against serogroups A, C, W, and Y:
  - o at baseline (Day 1, Month 0) and at 1 month after the first (Day 31, Month 1) and the last vaccination (Day 211, Month 7) for the ABCWY group, and
  - o at baseline (Day 1, Month 0) and 1 month after the single MenACWY vaccination for the ACWY group (Day 31, Month 1).
- The geometric mean titers (GMTs) against serogroups A, C, W, and Y:
  - o at baseline (Day 1, Month 0) and at 1 month after the first (Day 31, Month 1) and the last (Day 211, Month 7) vaccinations for the ABCWY group, and
  - o at baseline (Day 1, Month 0) and 1 month after the single MenACWY vaccination for the ACWY group (Day 31, Month 1).
- The geometric mean ratios (GMRs) against serogroups A, C, W, and Y:
  - o at 1 month after the first (Day 31, Month 1) and the last vaccination (Day 211, Month 7) for the ABCWY group as compared to baseline (Day 1, Month 0) and
  - o at 1 month after the MenACWY vaccination (Day 31, Month 1) for the ACWY group as compared to baseline (Day 1, Month 0).

The immune response to the MenABCWY vaccine (0,6-month schedule) against *N. meningitidis* serogroup B indicator strains, at pre-vaccination (Day 1, Month 0) and at 1 month after the **last** MenABCWY vaccination will be demonstrated for participants in the FAS (as defined in Section 5.4) from:

• The percentages of participants with hSBA titers ≥LLOQ for each and all serogroup B indicator strains at baseline (Day 1, Month 0) and at 1 month after the last vaccination (Day 211, Month 7) for the ABCWY group.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


- The percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers against each *N. meningitidis* serogroup B indicator strains at 1 month after the last vaccination (Day 211, Month 7) relative to baseline (Day 1, Month 0) for the ABCWY group.
- GMTs against each serogroup B indicator strains at baseline (Day 1, Month 0) and at 1 month after the last vaccination (Day 211, Month 7) for the ABCWY group.
- GMRs against each serogroup B indicator strains at 1 month after the last vaccination (Day 211, Month 7) as compared to the baseline (Day 1, Month 0) for the ABCWY group.



Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


ACWY group (Day 31, Month 1).

#### 2.5.4. PRIMARY SAFETY ENDPOINTS

The safety and reactogenicity of the MenABCWY and MenACWY vaccines will be demonstrated for participants in the corresponding Safety Sets (as defined in Sections 0, 5.6.2 and 5.6.3) from:

- The frequencies and percentages of participants with solicited administration site events (i.e., injection site pain, erythema, swelling, induration) and solicited systemic events (i.e., fever [body temperature ≥38.0°C/100.4°F], nausea, fatigue, myalgia, arthralgia, headache) during the 7 days (including the day of vaccination) following vaccination at Day 1, Month 0 (for the ABCWY and ACWY groups) and Day 181, Month 6 (for the ABCWY group).
- The frequencies and percentages of participants with any unsolicited AEs (including all SAEs, AEs leading to withdrawal, AESIs and medically attended AEs) during the 30 days (including the day of vaccination) following vaccination at Day 1, Month 0 (for the ABCWY and ACWY groups) and Day 181, Month 6 (for the ABCWY group).
- The percentages of participants with SAEs, AEs leading to withdrawal, AESIs and medically attended AEs throughout the study period (Month 0 to Month 12).

# 3. STUDY DESIGN

# 3.1. GENERAL DESCRIPTION

The study design diagram is provided in

Figure 1.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Figure 1 Study Design Overview



ACWY = *Menveo*; BS = blood sample; ESFU = extended safety follow-up; MenB = *Bexsero*; N = number of participants; T = telephone contact; V = visit

- Approximately 1206 participants will be randomized in a 1:1 ratio to achieve 1084 evaluable participants (at least 542 per group). Participants to receive:
  - ABCWY: At least 603 participants will receive 2 doses of the MenABCWY vaccine at

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C B4DEE6C228977964.docx


<sup>&</sup>lt;sup>a</sup> Bexsero is given for compliance with standard of care

<sup>&</sup>lt;sup>b</sup> Insufficient blood volume may lead to test cancellation and jeopardize the statistical power. Hence, every effort must be made to collect blood volume as per protocol requirements.

- Visit 1 (Day 1) and Visit 3 (Day 181) (0,6-month schedule) and 1 dose of placebo at Visit 4 (Day 211).
- ACWY: At least 603 participants will receive 1 dose of MenACWY vaccine at Visit 1 (Day 1) (single dose) and 2 doses of MenB vaccine at Visit 3 (Day 181) and Visit 4 (Day 211).

Randomization will be minimized for country. Study vaccine groups, intervention and blinding foreseen in the study are presented in

#### Figure 1 and

Table 1. For further details please refer to Section 3.0 of the protocol.

Table 1 Study Vaccine Groups, Intervention, and Blinding Foreseen in the Study

| Study<br>Vaccine<br>Group | Number of<br>Participants | Age<br>(Min to Max) | Intervention | Blinding |
|---|---|---|---|---|
| ADCWV | 625 | 15 to 25 years | MenABCWY | V1 to T5:<br>Observer-blind |
| ABCWY | 023 | 15 to 25 years | Placebo | |
| ACWY | 625 | 15 to 25 years | MenACWY | V1 to T5: |
| ACWI | 023 | 15 to 25 years | MenB | Observer-blind |

MenACWY = Menveo; MenB = Bexsero; T = telephone contact; V = visit

# 3.2. SCHEDULE OF EVENTS

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Schedule of events can be found in Section 1.3 of the protocol.

# 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

The visit window in the protocol is -5/+14 days for visits 2, 3 and 4. For the statistical analysis this window will be -7/+28 days for each visit.

There are no other changes to planned analyses in the protocol. However, during special circumstances such as the COVID-19 pandemic, the specific guidance from local public health and other competent authorities regarding the protection of individuals' welfare will be applied. For the duration of such special circumstances, some measures may impact the data and analysis:

- Delayed FPI
- Protocol deviations due to COVID-19
- Missed visits due to COVID-19
- Missed or modified assessments
- Treatment interruptions or delays
- Early study discontinuation or withdrawals due to having COVID-19 or COVID-19 related issues
- Adverse events or SAEs due to COVID-19

The number and percentage of participants experiencing any of the COVID related consequences listed above will be presented.

# 4. PLANNED ANALYSES

The following analyses will be performed for this study:

- Interim analysis
- Final Analysis

# 4.1. DATA MONITORING COMMITTEE (DMC)

There will be no DMC for this study.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


# 4.2. INTERIM ANALYSIS

An interim analysis of safety objectives will be conducted after at least 50% of participants have completed Visit 4. An interim analysis of immunological objectives may also be performed after all participants have completed Visit 4. If performed, the assessment of the primary immunological objectives will follow the order described in section 16.1.3 with analysis of family 1 preceding that of family 2.

The interim analysis will be performed by the unblinded analysis team who are independent of the blinded analysis team. Only unblinded analysis tables will be provided to avoid the reviewer being unblinded at a participant level.

# 4.3. FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics following GlaxoSmithKline authorization of this Statistical Analysis Plan, Database Lock, Sponsor Authorization of Analysis Sets and Unblinding of intervention.

# 5. ANALYSIS SETS

Agreement and authorization of participants included/excluded from each analysis set will be conducted prior to the unblinding of the study.

# 5.1. Process for Analysis Set Assignment

- Preliminary analysis sets will be derived, prior to the database lock, to the extent that data is available.
- Data listings presenting participants excluded from each preliminary analysis set and reasons
  for exclusion will be prepared for sponsor review ahead of database lock (during the data
  review meeting) in order to allow appropriate related data queries to be issued.
- The final analysis sets will be derived after database lock and will use the final study data, i.e., clinical database (CRF), external vendor data (serological results), eDiaries and protocol

 $\label{local-problem} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


- deviations log.
- Data listings presenting participants excluded from each final analysis set and reasons for exclusion will be prepared for sponsor review ahead of unblinding for a final review and approval.
- Customer authorization of the analysis sets will be necessary to unblind the data after database lock.

# **5.2.** ENROLLED SET [ENR]

The enrolled set (ENR) will contain all participants who agreed/participants for whom parent(s)/legally acceptable representative agreed to participate in a clinical study after completion of the informed consent process, who meet screening/eligibility criteria and randomized or received study intervention or undergone an invasive procedure.

For analyses and displays based on ENR, participants will be classified according to randomized intervention.

# 5.3. EXPOSED SET [ES]

The exposed set (ES) will contain all participants who received at least 1 dose of the study intervention.

The allocation in a group is done according to all administered interventions. If there is any doubt whether a participant was vaccinated or not, they will be assumed vaccinated for the purposes of analysis. Participants will be classified according to intervention received.

# 5.4. FULL ANALYSIS SET [FAS]

The FAS will contain all participants who received at least 1 dose of the study intervention and have post-vaccination immunogenicity data, i.e., available hSBA titer for at least one serogroup (A, B, C, W or Y).

For analyses and displays based on the FAS, participants will be classified according to the randomized intervention.

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


Note: The intent-to-treat principle is preserved, despite the exclusion of participants randomized who did not receive the study intervention, because the decision of whether or not to begin the intervention could not be influenced by knowledge of the assigned intervention, i.e. the study medication is blinded.

# 5.5. PER PROTOCOL ANALYSIS SET [PPS]

The PPS will contain all participants who received at least 1 dose of the study intervention to which they are randomized and have post-vaccination data (FAS) minus participants with protocol deviations that lead to exclusion from the PPS, as defined prior to analysis.

# 5.6. SAFETY ANALYSIS SETS

In case of a vaccination error (wrong vaccine), participants will be analyzed as "treated" (i.e., according to the vaccine a participant receives, rather than the vaccine to which the participant is randomized).

# 5.6.1. UNSOLICITED SAFETY ANALYSIS SET [USS]

The unsolicited safety analysis set (USS) will contain all participants who received at least 1 dose of the study intervention (ES) that report unsolicited AEs/report not having unsolicited AEs.

## 5.6.2. SOLICITED SAFETY ANALYSIS SET [SSS]

The solicited safety analysis set (SSS) will contain all participants who received at least 1 dose of the study intervention (ES) who have solicited safety data.

#### 5.6.3. OVERALL SAFETY ANALYSIS SET [OSS]

The overall safety analysis set (OSS) will contain all participants who are in the Solicited Safety Set and/or Unsolicited Safety Set.

# 5.7. OVERVIEW OF ANALYSIS BY PROTOCOL DEVIATION (PD)

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Details of PDs can be found in the Protocol Deviation Management Plan and in APPENDIX 3 of this SAP.

# 6. GENERAL CONSIDERATIONS

Immunogenicity and safety endpoints will be summarized descriptively (frequency and percent for categorical data; and number of participants with non-missing observations, mean [or geometric mean], standard deviation [SD] [or geometric standard deviation {GSD}], median, minimum, and maximum for continuous data, unless specified otherwise) at all relevant study visits, as appropriate. In summary tables for categorical data for which categories are defined on the electronic case report form (eCRF), all categories will be presented as specified, even if the participant count within that category is zero.

Unless otherwise specified, all data collected during the trial will be presented in the data listings.

# 6.1. REFERENCE START DATE AND STUDY DAY

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of the first dose of study medication, (Day 1 is the day of the first vaccination).

- If the date of the event is on or after the reference date then:
  - $\circ$  Study Day = (date of event reference date) + 1.

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the data listings.

## **6.2.** BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered pre-baseline, but Adverse Events (AEs)

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


and medications commencing on the reference start date will be considered post-baseline.

# 6.3. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

Not applicable.

# **6.4.** WINDOWING CONVENTIONS

The following table describes assignment of visit windows to the following data for purposes of the immunogenicity analysis:

Table 2 Visit Windows for Immunogenicity by Visit

| Assigned Study Day (Inclusive) | | Visit<br>Assigned | Day Assigned | Month Assigned |
|---|---|---|---|---|
| From | То | | | |
| 1 (pre-vaccination) | 1 (pre-vaccination) | Visit 1 | 1 | Baseline |
| 24 | 59 | Visit 2 | 31 | Month 1 |
| 173 | 208 | Visit 3 | 181 | Month 6 |
| 24* | 59* | Visit 4 | Visit 3 + 31 | Month 7 |

<sup>\*</sup> Based on number of days from visit 3

# **6.5.** STATISTICAL TESTS

The default significance level will be (5%); confidence intervals will be 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

# **6.6.** COMMON CALCULATIONS

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


#### **Geometric Mean Titer/Concentration (GMT/GMC)**

Distributions of antibodies are generally skewed to the right (Nauta, 2010). Therefore, prior to any statistical analysis that assumes normally distributed observations, antibody titers or concentrations will be  $log_{10}$ -transformed. GMTs [/GMCs] and their 95% CIs are computed by exponentiating (base 10) of the  $log_{10}$  titers.

The GMT [/GMC] will be calculated using the following formula:

$$10^{\left(\frac{\sum_{i=1}^{n}\log 10(t_i)}{n}\right)}$$

Where  $t_1, t_2, ..., t_n$  are *n* observed immunogenicity titers/concentrations.

#### Geometric Mean Ratio (GMR)

GMRs measure the changes in immunogenicity titers/concentrations within participants.

The GMR will be calculated using the following formula:

$$10^{\left(\frac{\sum_{i=1}^{n_g} \log 10^{(v_{ij}}/v_{ik})}{n_g}\right)} = 10^{\left(\frac{\sum_{i=1}^{n_g} \log 10(v_{ij}) - \log 10(v_{ik})}{n_g}\right)}$$

where, for  $n_g$  participants in vaccine groups g = 1 and 2,  $v_{ij}$  and  $v_{ik}$  are observed immunogenicity titers/concentrations for participant i at time-points j and k,  $j \neq k$ .

#### 4-fold rise

For the serogroups A, C, W, Y and for each of the serogroup B indicator strains evaluation the 4-fold rise is defined as:

- a post-vaccination hSBA titer ≥16 for participants with a pre-vaccination hSBA titer <4;
- a post-vaccination hSBA titer ≥4 times the LLOQ for participants with a pre vaccination hSBA titer ≥limit of detection (LOD) but <LLOQ; and,
- a post-vaccination hSBA titer ≥4 times the pre-vaccination titer for participants with a prevaccination hSBA titer ≥LLOQ.

B4DEE6C228977964.docx


# 6.7. SOFTWARE VERSION

All analyses will be conducted using SAS version 9.4 or higher.

## 7. STATISTICAL CONSIDERATIONS

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following covariates and factors will be used in the analyses in addition to the vaccine group. For details of their inclusion in the models, see the specific analysis subsections in Section 16.

- Baseline titers as a covariate in the Analysis of Covariance (ANCOVA) models
- Country as a factor in the Analysis of Variance (ANOVA) and ANCOVA models.

# 7.2. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers in approximately 4 countries. Randomization to vaccine group will be minimized by country. Additional analyses by country may be conducted as deemed necessary.

For continuous endpoints (GMT/GMR), the vaccine group effects will be investigated using a linear model that includes a factor for country differences but will not consider vaccine-by-country interaction, i.e., the model only considers effects for country and vaccine. If the statistical model does not converge due to the factor "country", a model without country effect will be fitted instead. If significant vaccine effects are found in a trial, there will be an exploration of the heterogeneity of vaccine group effects across countries. Results of vaccine by country interaction analysis will be provided in Appendix 16.1.9 of the Clinical Study Report (CSR).

# 7.3. MISSING DATA

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


There will only be limited imputation of missing data. To minimize the effect of dropouts and missing data, the study period will be divided into time intervals for statistical analysis of safety.

#### **Unsolicited Adverse Events Missing or Partial Dates**

Missing and partial AE start dates will be imputed as described in APPENDIX 2, only to determine the relationship between the start date of the event and the first dose date of vaccination. Partial dates will be presented as recorded in the data listings.

#### Missing intensity and relatedness for unsolicited AEs

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### **Missing Solicited Event Measurements**

On the solicited events eDiary, participants are instructed to enter a measurement for solicited administration site events (i.e., injection site pain, erythema, swelling, induration) and solicited systemic events (i.e., fever [body temperature  $\geq 38.0^{\circ}$ C/100.4°F], nausea, fatigue, myalgia, arthralgia, headache) during the 7 days (including the day of vaccination) following vaccination at Day 1, Month 0 and Day 181, Month 6.

#### Titers Measured Below (or Above) the LLOQ (or ULOQ)

For the hSBA assay, a titer value measured below LLOQ will be imputed to a value that equal to LLOQ/2 in summaries and analyses but will be listed as reported in the raw serology data. For example, a serologic assay with LLOQ = 30 generally reports values below LLOQ as "<30". The data listings will present the values as "<30", while values of 15 are to be used in the summaries and analyses.

Titer values measured as above ULOQ will be imputed at the ULOQ value.

Otherwise, missing immunogenicity values are considered Missing Completely at Random (MCAR) and "therefore will not contain information that impact the result of the analysis (i.e., not informative). Imputation methods will therefore not be used.

# 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


For the multiplicity adjustment, all hypotheses will be ranked into two families, family 1 and family 2. Fixed sequential testing with full alpha propagation in these pre-ordered hypotheses families will be applied. Refer protocol section 9.2 sample size determination for more details.

# 7.5. ACTIVE-CONTROL STUDIES INTENDED TO SHOW NON-INFERIORITY

NI will be demonstrated if, the lower limit of 2-sided 95% confidence interval (CI) for the percent difference in 4-fold rise (refer to Section 6.6) in hSBA titers (p\_MenABCWY- p\_MenACWY) is above -10%, for each N. meningitidis A, C, W, and Y serogroup. Additional details provided in Section 16 of this SAP.

# 7.6. EXAMINATION OF SUBGROUPS

Subgroup analyses will be conducted for the Primary immunogenicity analyses only. It should be noted that the study was not designed to detect treatment differences with high statistical power within subgroups. The following subgroups will be assessed and described within the immunogenicity analysis sections: Gender (Female, Male), Race (White, Non-white), Age in years (15 to <18,  $\ge$ 18-25), Country (by country, and 'US vs. Rest of the World (ROW)'.

# 7.7. RANDOMIZATION AND BLINDING

#### 7.7.1. METHOD OF GROUP ASSIGNMENT AND RANDOMIZATION

For further details please refer to Section 6.3 of the protocol.

#### 7.7.2. DEFINITION OF RANDOMIZATION/VACCINATION ERRORS

The list below provides some examples of potential errors that may occur during vaccination:

- Administration of concomitant vaccine(s) forbidden in the protocol (code 1040)
- Randomisation failure (participant not randomized in correct group) (code 1050)
- Randomisation code was broken (code 1060)

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


- Dosing not according to protocol (code 1070)
- Dosing after a Temperature deviation (code 1080)
- Dosing after expiration (code 1090)

Randomization errors will be summarized by presenting the number and percentage of participants with randomization errors for the enrolled set. Participants with randomization errors should be analyzed as randomized in FAS, excluded from PPS and analyzed as received for Safety.

# 8. OUTPUT PRESENTATIONS

Programming Conventions for Outputs shows conventions for presentation of data in outputs.

The templates (table shells) provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and data listings to be provided by IQVIA Biostatistics.

Statistical output numbering will follow 'ICH E3 Structure and Content of Clinical Study Reports'.

# 9. DISPOSITION AND WITHDRAWALS

All participants from the ENR Set will be accounted for in this study.

# 9.1. DISPOSITION

The number of enrolled, vaccinated (at least 1 vaccination, full vaccination course), completed participants, screening failures, reason for withdrawal, and reason for exclusion from analysis sets, as well as number of participants in FAS and PPS will be reported by group for the ENR set. Additionally, the number of participants discontinuing the study and the reason for discontinuation, including COVID-19, will be presented.

A data listing of the disposition information will be provided. If applicable, early study discontinuation or withdrawals due to having COVID-19 or COVID-19 related issues will be presented. The number of

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


participants who discontinued study drug and who withdrew from the Study due to COVID-19 infection or issues related to the COVID-19 pandemic will be presented.

# 9.2. PROTOCOL DEVIATIONS

Protocol deviations will be collected in a PD log, as detailed in the Protocol Deviations Management Plan.

All protocol deviations will be assessed as important or non-important. Protocol deviations will be reviewed by the GSK Team, and their status confirmed by the time that all data are cleaned for the Final Analysis. APPENDIX 3 lists PDs that affect the validity of the immunogenicity measurements and result in exclusion of participants from the PPS.

A summary presenting the number and percentage of participants in each PD category will be presented for participants in the ENR set, by vaccine group and overall, and a data listing will be provided for participants with protocol deviations during the study. Additionally, a data listing of PDs for participants who are excluded from the PPS will be generated.

A summary presenting the number and percentage of participants with a protocol deviation related to COVID-19 in each PD category will be presented for participants in the ENR set, by vaccine group and overall. Additionally, PDs related to COVID-19 will be flagged in the PD listing.

# 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the ENR, ES, FAS and PPS. No statistical testing will be carried out for demographic or other baseline characteristics.

The following demographic and other baseline characteristics will be reported for this study: Age (years) at the time of the first vaccination, Sex, Race, Ethnicity, Weight (kg), Height (cm) and Body Mass Index (BMI) (kg/m²). Descriptive statistics (mean, standard deviation [SD], median, minimum and maximum) for age, height, weight, and body mass index will be calculated overall and by vaccine group. Distributions of participants by sex, race, and ethnic origin will be summarized overall and by vaccine group.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


## 10.1. DERIVATIONS

#### Age (years) at first vaccination

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

- DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years
- DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

Note: If we have partial DOB, the DOB will be imputed as described in APPENDIX 2.

#### Weight

Weight will be presented in kilograms. Weights reported in pounds will be converted as follows:

• Weight in kilograms = Weight in pounds / 2.2

#### Height

Height will be presented in centimeters. Heights reported in feet and inches will be converted as follows:

• Height in centimeters = Height in inches x 2.54

#### **Body mass index (BMI)**

BMI will be calculated as follows:

• BMI (kg/ $m^2$ )= (Weight in kilograms) / (Height in meters)<sup>2</sup>

## **Temperature**

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

• Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

# 11. VACCINATION AND MEDICAL HISTORY

Vaccination and Medical History information will be presented for the ES.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


- Vaccination History:
  - Identity of the primary MenACWY vaccination
  - o Age at primary MenACWY vaccination.
- Medical History will be coded using the current version of the Medical Dictionary for Regulatory Activities (MedDRA):
  - Medical History conditions are defined as those conditions which stop prior to or at the first vaccination.
  - o Presented by System Organ Class (SOC) and Preferred term (PT).

# 12. CONCOMITANT ILLNESSES

Concomitant Illnesses (also captured on the Medical History page) will be presented for the ES.

- Concomitant Illnesses will be coded using the current version of the MedDRA dictionary:
  - Concomitant Illnesses are conditions which started prior to the first vaccination and are ongoing at the first vaccination.
  - o Presented by SOC and PT.

# 13. MEDICATIONS

Medications will be presented for the ES and coded using the current version of World Health Organization (WHO) Drug dictionary. Medications will be presented by anatomical therapeutic chemical (ATC) classification and preferred drug name, overall and by vaccine group.

See APPENDIX 2 for handling of partial dates for medications, in the case where it is not possible to define a medication as prior or concomitant, the medication will be classified by the worst case; i.e. concomitant.

- 'Prior' medications are medications which started and stopped prior to the first vaccination.
- 'Concomitant' medications are medications which:
  - o started prior to, on or after the first vaccination, AND

 $\label{local-converter-lamb-conver$ 

B4DEE6C228977964.docx


o ended on or after the date of first vaccination or were ongoing at the end of the study.

# 14. STUDY MEDICATION EXPOSURE

The total time in the study (including follow-up after the last vaccination) will be summarized as a continuous variable by vaccine group and overall. The total time in study is defined as the number of days from the first vaccination to the date of last contact specified on the End of Study Visits form. This will generally be the date of the last telephone contact (scheduled on Day 361). The vaccination date/time information will be listed for each participant.

# 14.1. DERIVATIONS

Total time in study (days) = date of last contact – date of first vaccination + 1.

# 15. STUDY MEDICATION COMPLIANCE

Compliance to study medication will be presented for the ES.

The number and percentage of participants receiving 1 dose, 2 doses or all 3 doses will be presented overall and by vaccine group for the ES. For each intervention, the number of participants receiving the vaccine outside the specified window will be presented.

The number and percentage of participants who missed each dose or received the dose outside the planned window due to COVID-19 will be presented (if applicable) overall and by vaccine group for the ES.

# 16. IMMUNOGENICITY OUTCOMES

# 16.1. PRIMARY IMMUNOGENICITY

#### 16.1.1. Primary Immunogenicity Variable & Derivations

The first co-primary immunogenicity variable is the percentages of participants with a 4-fold rise (refer to

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Section 6.6) in hSBA titers against N. meningitidis serogroups A, C, W, and Y at 1 month after the **second** vaccination for the ABCWY group (Day 31, Month 1), and 1 month after the single dose of MenACWY vaccination for the ACWY group (Day 31, Month 1), relative to baseline (Day 1, Month 0).

The second co-primary immunogenicity variable is the percentages of participants with a 4-fold rise (refer to Section 6.6) in hSBA titers against N. meningitidis serogroups A, C, W, and Y at 1 month after the **first** vaccination for the ABCWY group (Day 31, Month 1), and 1 month after the single dose of MenACWY vaccination for the ACWY group (Day 31, Month 1), relative to baseline (Day 1, Month 0).

## 16.1.2. MISSING DATA METHODS FOR PRIMARY IMMUNOGENICITY VARIABLE(S)

Refer to Section 7.3.

#### 16.1.3. PRIMARY ANALYSIS OF PRIMARY IMMONOGENICITY VARIABLE

The following study hypotheses are ordered into 2 families that will be tested in sequential design with full alpha propagation. Family 1 will be tested first and family 2 will only be tested if the hypothesis in family one is successfully demonstrated.

First Co-Primary Immunogenicity Objective (Family 1):

The first co-primary immunogenicity objective is to demonstrate the immunological non-inferiority of the antibody response to MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with MenACWY, as measured by percentage of participants with 4-fold rise (refer to Section 6.6) in hSBA titer against each of the *N. meningitidis* serogroups A, C, W, and Y, at 1 month after the **second** MenABCWY vaccination and 1 month after the MenACWY vaccination (single dose). This translates to the following hypotheses:

 $H_0$ : (p1 MenABCWY<sub>(i)</sub> - p1 MenACWY<sub>(i)</sub>)  $\leq -10\%$ 

VS.

 $H_1$ : (p1 MenABCWY<sub>(i)</sub> - p1 MenACWY<sub>(i)</sub>) > -10%

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Where p1\_MenABCWY<sub>(i)</sub> denotes the percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers for serogroups i=A, C, W, and Y, 1 month after the **second** vaccination of MenABCWY group and p1\_MenACWY<sub>(i)</sub> denotes the percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers for serogroups i=A, C, W, and Y, 1 month after the single vaccination of MenACWY group.

The primary immunogenicity analysis will be performed for the PPS. The primary immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine, will be demonstrated if the lower limit (LL) of the 2-sided 95% CI for the group difference in percentages of participants achieving a 4-fold rise (refer to Section 6.6) in hSBA titers is above -10%, for each serogroup.

For each of the serogroups A, C, W, Y the percentages of participants with 4-fold rise (refer to Section 6.6), and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method (Clopper and Pearson, 1934) will be calculated for each vaccine group at 1 month post **second** vaccination. The standardized asymptotic CIs between group differences in percentages will be derived using the method of Miettinen and Nurminen (Nurminen, 1985).

Second Co-Primary Immunogenicity Objective (Family 2):

The second co- primary immunogenicity objective is to demonstrate the immunological NI of the antibody response to MenABCWY vaccine, compared to MenACWY vaccine given to healthy participants, previously primed with MenACWY, as measured by percentage of participants with 4-fold rise (refer to Section 6.6) in hSBA titer against each of the *N. meningitidis* serogroups A, C, W, and Y, at 1 month after the **first** MenABCWY vaccination and 1 month after the MenACWY vaccination (single dose). This translates to the following hypotheses:

 $H_0$ :  $(p2\_MenABCWY_{(i)} - p2\_MenACWY_{(i)}) \le -10\%$ 

VS.

 $H_1$ : (p2 MenABCWY<sub>(i)</sub> – p2 MenACWY<sub>(i)</sub>) > -10%

Where p2\_MenABCWY<sub>(i)</sub> denotes the percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers for serogroups i=A, C, W, and Y, 1 month after the **first** vaccination of MenABCWY group

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx

and p2\_MenACWY<sub>(i)</sub> denotes the percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers for serogroups i=A, C, W, and Y, 1 month after the single vaccination of MenACWY group.

The secondary immunological non-inferiority of the MenABCWY vaccine, compared to MenACWY vaccine, will be demonstrated if the lower limit (LL) of the 2-sided 95% CI for the group difference in percentages of participants achieving a 4-fold rise (refer to Section 6.6) in hSBA titers is above -10%, for each serogroup

For each of the serogroups A, C, W, Y the percentages of participants with 4-fold rise (refer to Section 6.6), and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method (Clopper, 1934) will be calculated for each vaccine group, at 1 month after the **first** vaccination for the ABCWY group (Day 211, Month 7), and 1 month after the single dose of MenACWY vaccination for the ACWY group (Day 31, Month 1). The standardized asymptotic CIs between group differences in percentages will be derived using the method of Miettinen and Nurminen (Nurminen, 1985). The secondary immunological non-inferiority analysis will be performed for the PPS.

# 16.1.4. SENSITIVITY ANALYSIS OF PRIMARY IMMUNOGENICITY VARIABLE(S)

Each co-primary immunogenicity objective will be analysed as a sensitivity analysis using a logistic regression with margins calculated by Taylors approximation with the minimization factors as covariables.

### 16.1.5. SUBGROUP ANALYSIS OF PRIMARY IMMUNOGENICITY VARIABLE(S)

The primary immunogenicity variables will be analysed for subgroups listed in Section 7.6

# 16.2. SECONDARY IMMUNOGENICITY

The secondary immunogenicity analyses will be performed for the FAS.

### 16.2.1. SECONDARY IMMUNOGENICITY VARIABLES & DERIVATIONS

16.2.1.1. Immune Response, Serogroups A, C, W and Y (measured by hSBA)

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


The immune response to MenABCWY (0,6-month schedule) and MenACWY (single dose) vaccines against *N. meningitidis* serogroups A, C, W, and Y, at pre-vaccination (Day 1, Month 0) and 1 month after the **first and last** MenABCWY vaccinations and 1 month after the single MenACWY vaccination will be demonstrated using:

- Logarithmically transformed (base 10) hSBA titers and percentages of participants with hSBA titers
   >LLOO:
  - o at baseline (Day 1, Month 0) and at 1 month after the first (Day 31, Month 1) and the last vaccination (Day 211, Month 7) for the ABCWY group, and
  - o at baseline (Day 1, Month 0) and 1 month after the single MenACWY vaccination for the ACWY group (Day 31, Month 1).

# 16.2.1.2. Immune Response, Serogroup B Indicator Strains (measured by hSBA)

The immune response to the MenABCWY vaccine (0,6-month schedule) against *N. meningitidis* serogroup B indicator strains:

- M14459 for factor H binding protein [fHbp] antigen
- M13520 for NHBA antigen
- 96217 for Nad A antigen; and
- NZ98/254 for PorA P1.4 antigen

will be demonstrated using:

- Logarithmically transformed (base 10) hSBA titers
- The percentages of participants with hSBA titers ≥LLOQ for each and all serogroup B indicator strains at baseline (Day 1, Month 0) and at 1 month after the last vaccination (Day 211, Month 7) for the ABCWY group. For the 'all' serogroup B indicator strains to be considered as satisfying the '≥LLOQ' criteria, all 4 of the serogroup indicator strains hSBA titers must be ≥LLOQ.
- The percentages of participants with 4-fold rise (refer to Section 6.6) in hSBA titers against each *N. meningitidis* serogroup B indicator strains at 1 month after the last vaccination (Day 211, Month 7) relative to baseline (Day 1, Month 0) for the ABCWY group.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


#### 16.2.2. MISSING DATA METHODS FOR SECONDARY IMMONOGENICITY VARIABLES

Refer to Section 7.3

#### 16.2.3. ANALYSIS OF SECONDARY IMMUNOGENICITY VARIABLES

16.2.3.1. Immune Response Analysis, Serogroups A, C, W and Y (measured by hSBA)

For each of the 4 *N. meningitidis* serogroups A, C, W, and Y the percentages of participants with hSBA titers ≥LLOQ and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method (Clopper) will be calculated at baseline (Day 1, Month 0), and at 1 month after the **first** (Day 31, Month 1) and the **last** vaccination (Day 211, Month 7) for the ABCWY group, and at baseline (Day 1, Month 0) and 1 month after the single MenACWY vaccination for the ACWY group (Day 31, Month 1).

The titers at baseline (Day 1, Month 0), at 1 month after the **first** (Day 31, Month 1) and the **last** vaccination (Day 211, Month 7) for the ABCWY group, and at 1 month after the single MenACWY vaccination (Day 31, Month 1) in the ACWY group, will be logarithmically transformed (base 10) to fulfill the normal distribution assumption.

GMTs and 95% CIs will be calculated by exponentiating (base 10) the least squares means and the lower and upper limits of the 95% CIs of the log-transformed titers (base 10) obtained from:

- an ANOVA with factors for vaccine group and country.
- an ANCOVA with baseline titers as a covariate, and factors for vaccine group and country.

GMRs (post vaccination/baseline titer) and associated 2-sided 95% CIs will be computed for each group and for each serogroup at each visit. GMRs will be calculated by exponentiating (base 10) the least squares means and the lower and upper limits of the 95% CIs of the log-transformed titers (base 10) obtained from an ANOVA with factors for vaccine group and country.

Additionally, GMTs and GMRs group ratios between the 2 vaccine groups and their respective 95% CIs will be computed by exponentiating the difference of the least square means of the log-transformed titers and the lower and upper limits of the 95% CIs on the difference obtained from the ANOVA model above.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


#### 16.2.3.2. Immune Response Analysis, Serogroup B Indicator Strains (measured by hSBA)

For *N. meningitidis* B indicator strains (M14459 for factor H binding protein [fHbp] antigen, M13520 for NHBA antigen, 96217 for NadA antigen and NZ98/254 for PorA P1.4 antigen):

- the percentages of participants with hSBA titers ≥LLOQ for each and all serogroup B indicator strains, and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method (Clopper) will be calculated for the MenABCWY vaccine group at at baseline (Day 1, Month 0), and at 1 month after the **last** vaccination (Day 211, Month 7).;and
- the percentage of participants with 4-fold rise (refer to Section 6.6) relative to baseline for each serogroup B indicator strains, and the corresponding exact 2-sided 95% CIs based on Clopper-Pearson method (Clopper) will be calculated for the MenABCWY vaccine group at at 1 month after the **last** vaccination (Day 211, Month 7).

GMTs and associated 2-sided 95% CIs will be computed for each serogroup B indicator strain at baseline (Day 1, Month 0), and at 1 month after the **last** vaccination (Day 211, Month 7) for the ABCWY vaccine group. The hSBA titers at baseline (Day 1, Month 0), and the hSBA titers at 1 month after the last vaccination (Day 211, Month 7) for the ABCWY group, will be logarithmically transformed (base 10) to fulfill the normal distribution assumption. For each *N. meningitidis* B test strain (M14459, M13520, 96217 and NZ98/254), the GMTs pre- and post-vaccination with their 95% CIs will be calculated by exponentiating (base 10) the means and the lower and upper limits of the 95% CIs of the log-transformed titers (base 10) values.

GMRs (post-vaccination/baseline titer) and associated 2-sided 95% CIs will be computed for each serogroup B indicator strain at 1 month after the **last** vaccination (Day 211, Month 7) for the ABCWY vaccine group, by exponentiating the corresponding log-transformed mean and 95% CI.



 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


Final 5.0

05SEP2022

Version Number:

**CONFIDENTIAL** Version Date:



Author:

PPD

Statistical Analysis Plan




Document:

Final 5.0 Author: Version Number: PPD



# 17. SAFETY OUTCOMES

The analysis of safety assessments in this study will include summaries of the following categories of safety data collected for each participant:

- Solicited administration site and systemic adverse events and indicators of solicited events.
- Unsolicited adverse events.

There will be no statistical comparisons between the vaccine groups for safety data, unless otherwise specified with the relevant section.

# 17.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded using the current version of the MedDRA dictionary.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


See APPENDIX 2 for handling of partial dates for AEs. In the case where it is not possible to determine if an AE started after the first vaccination or not, the AE will be considered to have started after the vaccination.

#### 17.1.1. SAFETY COMPLETENESS ANALYSIS

#### Solicited events (solicited administration site events and solicited systemic events)

The safety completeness analysis on solicited events aims to identify participants who completed the eDiary, irrespective of severity. The analysis will show the number of participants with valid data by solicited event, for each vaccination.

Four summaries will be produced:

- The frequencies of participants who provide eDiary information by vaccine group.
- For each solicited event, the frequencies of participants with valid data will be presented by vaccine group and time point: Day 1, Days 2, 3, 4, 5, 6 and 7.
- For each type of solicited event (administration site, systemic), the frequencies of participants with valid data by vaccine group, aggregated over time points: Day 1 Day 7.
- For each solicited event, the frequencies of participants with valid data by vaccine group, aggregated over time points: Day 1 Day 7.

For the corresponding percentages, the denominator will be the respective numbers of exposed participants, i.e., participants who received a vaccination and were still in-study for that time point or time interval, irrespective of whether an eDiary was available or not. All analyses will be based on the ES.

#### 17.1.2. SOLICITED EVENTS

For details please refer to Appendix 4 of the protocol. Solicited events will be summarized using the SSS.

Only solicited administration site (i.e., injection site pain, erythema, swelling, induration) and systemic (i.e., fever [temperature  $\geq$ 38.0°C/100.4°F], nausea, fatigue, myalgia, arthralgia, headache) adverse events reported in the diary card will be analyzed.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Solicited events will be reported daily starting on Day 1 and until Day 7 after each vaccination a Day 1 and Day 181 using structured eDiaries, i.e. Day 1 to Day 7 and Day 181 to 187. The analyses of solicited events will be done based on three intervals after each vaccination: Day 1 - 3, Day 4 - 7 and Day 1 - Day 7. Solicited site administration or systemic adverse events extending beyond 7 days will be presented separately. In addition:

- A solicited administration site or systemic adverse event ongoing after 7 days following each vaccination; or
- A solicited administration site or systemic adverse event that leads to a visit to a healthcare provider (medically attended AE); or
- A solicited administration site or systemic adverse event leading to the participant withdrawing from the study or the participant being withdrawn from the study by the investigator (AE leading to withdrawal); or
- A solicited administration site or systemic adverse event that otherwise meets the definition of an SAE
- Will be recorded and presented as an unsolicited AE.

For erythema, swelling and induration, recorded originally as diameters (mm), the following categorization will be used to summarize the data:

- None (< 25 mm) vs. any (>= 25 mm)
- None (< 25 mm), Mild (25-50 mm), Moderate (51-100 mm) and Severe (>100 mm)

Body temperature will be broken down by route of measurement according to the recommendations of the Brighton collaboration (<a href="www.brightoncollaboration.org">www.brightoncollaboration.org</a>) and will be summarized according to the 3 schemes described below:

• by 1.0 °C increments:

< 36.0

0 36.0 - 36.9

0 37.0 - 37.9

 $\label{local-problem} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


- 0 38.0 38.9
- 39.0 39.9
- o ≥40.0°
- $<38.0, \ge 38.0$  °C (i.e., 'no fever' versus 'fever')

Fever, defined as a body temperature of  $\geq 38^{\circ}$ C irrespective of route of measurement, will be integrated to the summaries as a systemic AE.

The analyses will encompass summaries of the data on five levels:

- 1. Daily reports of participants with solicited events.
- 2. Time of first onset of solicited events.
- 3. Solicited events, maximum event severity (i.e., severity grading scale as defined in Appendix 4 of the protocol) by event and interval Day 1 3, Day 4 7, and Day 1 7.
- 4. Duration of solicited events, excluding ongoing solicited events after Day 7.
- 5. Solicited events and indicators of solicited events, occurrence of at least one event by category (administration site, systemic) and interval Day 1 3, Day 4 7, Day 1 7 and extending beyond Day 7.

For studies using electronic diaries for the collection of solicited vents, a solicited event will be considered present only when a daily recording of grade 1 or more is present. For each of the time points or time intervals presented in the summaries, only participants with at least one observation for the solicited events in the interval of interest will be considered.

The analysis of solicited events after first vaccination will be reported separately from the analyses of solicited events after second vaccination. When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs

Level 1: Daily reports of solicited events

For each of the time points, only participants with at least one observation for the solicited events in the

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Statistical Analysis Plan


interval of interest will be considered. Data collected will be summarized (frequencies and percentages of participants) by vaccine group, solicited events, vaccination number and time point.

Level 2: Time of first onset of solicited events

The time of first onset is defined, for each participant, for each solicited event, as the time point at which the respective solicited event first occurred. For erythema, swelling and induration the following threshold will be used  $\geq 25$  mm. The summary will provide the frequencies and percentages of participants with first onset of each solicited events by vaccine group and vaccination number, and by each time point. For each vaccination the first onset of the AE will be used for each participant. For any vaccination the worst AE across all vaccinations per time point will be used. Note, 'not done' is treated identical to 'missing'.

Level 3: Solicited events, maximum event severity by event and interval

The maximum event severity will be defined if there is at least one non-missing observation within this time interval, each participant's data will be aggregated across the time points of the interval and summarized according to the maximal severity observed for each adverse event, followed by a summary across participants for each vaccine group and vaccination. Participants without any solicited events in the interval, i.e., missing values at each of the requested time points, will be removed from the denominator.

Level 4: Number of days with solicited events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The number of days with the AE is defined irrespective of severity. This means at least 'mild' solicited events that are assessed qualitatively  $\geq 25$ , mm for erythema, swelling and induration. If a solicited event continues beyond Day 7 the period after Day 7 is not added.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


The frequency distribution of the number of days will be provided in a summary table by vaccine group and vaccination, and by AE.

Level 5: Solicited events, occurrence of at least one event by category (administration site, systemic) and interval.

The occurrence of at least one solicited event is defined as "any" for a participant if he/she reports greater than "none" ≥ 25 mm, for erythema, swelling and induration for the respective event and "none" otherwise. The occurrence of at least one solicited event (i.e., none versus any) will be summarized by category (i.e., administration site, systemic, any), by vaccine group, by vaccination (after each vaccination and after any vaccination) and by time interval.

Use of antipyretics and analgesics to treat or prevent pain or fever will be summarized by frequencies and percentages of participants reporting use of the medications by type of use (prophylactic versus treatment) and for Day 1 - Day 3, Day 4 - 7, Day 1 - Day 7.

#### 17.1.3. UNSOLICITED ADVERSE EVENTS

The unsolicited AEs will be summarized per the USS.

All the unsolicited AEs occurring during the study, judged either as probably related, possibly related, or not related to vaccination by the investigator, will be recorded. The original verbatim terms used by investigators to identify adverse events in the CRFs will be mapped to preferred terms using the MedDRA dictionary. The unsolicited AEs will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. AEs judged by the investigator as at least possibly related to study vaccine will be summarized by vaccine group, according to system organ class and preferred term within system organ class. When an unsolicited AE occurs more than once for a participant, the maximal severity and strongest relationship to the vaccine group will be counted.

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an adverse event is between the first vaccination and the second vaccination, the relative dose will be the first vaccination.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

If an adverse event start date is missing or unknown, the AE will be considered as to have started after the first vaccination. For partially available dates, refer to APPENDIX 2.

Only adverse events with a start date on or after the first vaccination will be analyzed, i.e., excluding those after a participant has given informed consent but before the first vaccination. The selection of unsolicited AEs and the assignment to time intervals will be done by day of onset and not by days ongoing/persisting. AEs starting prior to the first vaccination, if any, will only be listed.

For each of the following intervals any unsolicited AE will be summarized:

- after each vaccination (from Day 1 to Day 31 and from Day 181 to Day 211, separately)
- after any vaccination (Day 1-31 and Day 181-211):
- entire study (Day 1 to end of study)

The following unsolicited adverse events will be summarized during the entire study:

- Possibly or probably related unsolicited AEs.
- Unsolicited AEs leading to death will be listed.
- Serious adverse events (SAEs).
- Possibly or probably related SAE.
- Possibly or probably related SAE leading to death
- Unsolicited AEs leading to premature withdrawal from study.
- Unsolicited AEs leading to discontinuation or delay in study vaccination.
- Unsolicited adverse events of special interest (AESI), as recorded on the Expedited AE report.
- Medically attended AEs.

 $\label{local-converter-app} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


Note: All the information required for the unsolicited AE summaries, including AESIs and medically attended AEs will be collected on the eCRF AE Form. Solicited events starting more than 7 days after the vaccination will also be considered as unsolicited AEs.

#### 17.1.4. COMBINED SOLICITED AND UNSOLICITED ADVERSE EVENTS

A summary of participants with all combined solicited events (regardless of their duration; where erythema, swelling and induration are reported as any events with a diameter >= 1 mm) and unsolicited AEs will be provided. Unsolicited events will be coded by MedDRA. For clintrial gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-SAEs will be produced by System Organ Class and according to occurrence of each event. For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages. Multiple events with the same preferred term which start on the same day are counted as only one occurrence. A further differentiation of combined AEs according to seriousness, severity, or relationship is not performed.

#### **17.1.5. COVID-19 EVENTS**

For the duration of special circumstances such as the COVID-19 pandemic, additional specific information will be summarized for the exposed set by vaccine group:

- Number of participants suspected, probable or confirmed for COVID-19 infection across diagnosis,
- Number of participants who had a COVID-19 diagnosis test and assessment performed
- Number of participants with positive, negative, or indeterminate results
- Incidence of COVID-19 reported as an adverse event or serious adverse event,
- Incidence of treatment discontinuation due to adverse event of COVID-19 infection,
- Incidence of adverse events over the time course of the trial (pre, during and post pandemic),
- Incidence of adverse by country or analysis region, age and gender over the time course of the trial (pre, during and post pandemic)

# 17.2. LABORATORY EVALUATIONS

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


A urine pregnancy test will be conducted as needed for women of childbearing potential. Pregnancy test results will be presented in a data listing.

# 18. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

Comments

These domains and/or variables will not be summarized or presented, but will be available in the clinical study database, SDTM and/or ADaM datasets.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


# 19. REFERENCES

Clopper CJ, Pearson ES. The use of confidential or fiducial limits illustrated in the case of the binomial. Biometrika 1934; 26:404-413.

Miettinen O., Nurminen M. Comparative analysis of 2 rates. Statistics in Medicine 1985; 4(2):213-26

Nauta J. Statistics in Clinical Vaccine Trials. 2010. Heidelberg: Springer.

U.S. Department of Health and Human Services, Food and Drug Administration, CDER/CBER (2016): Guidance for Industry Non-Inferiority Clinical Trials to Establish Effectiveness

ICH Harmonized Guideline for Estimands and Sensitivity Analysis in Clinical Trials E9 (R1). 2017.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


# APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

#### **IQVIA Output Conventions**

Outputs will be presented according to the IQVIA output conventions.

#### **Document Headers**

All TFL is to include the following header:

**GSK Vaccines** 

Vaccine: MenABCWY

Study 213171 (MenABCWY-19) - DELIVERY DESIGNATION

where delivery designation is the name of the current delivery, e.g., DRY-RUN, FINAL REPORT, etc.

#### **Dates & Times**

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

# **Spelling Format**

English US.

#### **Presentation of Vaccine Groups**

For outputs, vaccine groups will be represented as follows and in the given order:

| Vaccine Group | For Tables, Listings and Figures |
|---------------|----------------------------------|
| ABCWY | ABCWY + Placebo |
| ACWY | ACWY + Men B |

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


#### **Presentation of Visits**

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|----------------------------|------------|
| Baseline | BL |
| Day 1, Month 0 (Visit 1) | D1 (M0) |
| Day 31, Month 1 (Visit 2) | D31 (M1) |
| Day 181, Month 6 (Visit 3) | D181 (M6) |
| Day 211, Month 7 (Visit 4) | D211 (M7) |
| End of Study | EoS |

#### **Tables**

The 'Missing' category, when appropriate, will only be presented if participants qualify for this category. Otherwise, the row for 'Missing' will not be presented.

#### **Decimal places**

Decimal places for percentages and their corresponding confidence limits will be displayed with:

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 participants in each tabulated group
- one decimal when there are at least 50 participants in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of participants per tabulated group.
- O Differences in percentages and their corresponding confidence limits will be displayed with one more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with one decimal will be displayed with two decimals.

Decimal places for Demographic and baseline characteristics will be as follows:

- The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal.
- The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.
- The maxima and minima of transformed height variables will be displayed with no decimals.
- The maxima and minima of transformed weight variables will be displayed with no decimals

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C B4DEE6C228977964.docx


with the exception of values are below 10kg where one decimal will be displayed.

 The maximum and minima of transformed body temperatures will be displayed with one decimal.

#### **Serological Summary Statistics**

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

#### **Data Listings**

All data listings will be ordered by the following (unless otherwise indicated in the template):

- Randomized vaccine group (or intervention received if it's a safety output),
- Center-participant ID,
- Date (where applicable),
- For data listings where non-randomized participants would be included, these will appear in a category after the randomized vaccine groups labeled 'Not Randomized'.

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


#### **File Naming Convention**

The output files and corresponding SAS programs will have the same name.

The filename will start with 't', 'l' or 'f', respectively for table, listing or figure.

The filename will end with a brief description of the output content.

For output filenames (and corresponding SAS programs) that include numbers, include leading zeroes ('0') when the number is smaller than 10.

Elements in the file name will be separated by underscores '\_'.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


# APPENDIX 2. Partial Date Conventions

Imputed dates will NOT be presented in the data listings.

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30th.

The following exceptions apply:

- Imputed adverse event end date occuring before the actual start date
  - o If the imputed event end date occurs before the event start date then the imputed end date will be December 31<sup>st</sup>, unless this occurs after the study conclusion date in which case the earlier date is used.
- Adverse event start dates with missing day:
  - o If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month:
  - o If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

 $\label{local-converter-lambda} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


o Adverse event start dates with missing day and month:

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


# APPENDIX 3. PROTOCOL DEVIATIONS AND EXCLUSIONS FROM ANALYSIS SETS

Details of exclusions from each analysis sets are provided below. A complete list of participants excluded from each analysis set will be reviewed and confirmed by the sponsor prior to unblinding.

#### **Exclusion from Exposed Set (ES)**

'Study intervention not administered at all', 'Fraudulent data' and code 'Invalid informed consent or fraudulent data' will be used for identifying participants excluded from ES.

#### Exclusion from unsolicited and solicited safety set

#### **Unsolicited safety set**

'Study intervention not administered at all', 'fraudulent data', 'invalid informed consent' and 'no post-dose safety data' will be used for identifying participants excluded from the unsolicited safety set.

#### Solicited safety set

'Study intervention not administered at all', 'fraudulent data' and 'invalid informed consent' and 'no post-dose solicited safety data' will be used for identifying participants excluded from the solicited safety set.

 $\label{lem:lem:loc_converter} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


#### **Exclusion from Full Analysis Set (FAS)**

'Study intervention not administered at all', missing laboratory (Immunology) assessment (missed visit, blood draw not done at visit, sample not available for testing, result not available) and 'Fraudulent data' will be used for identifying participants excluded from the FAS.

# **Exclusion from Per-protocol analysis Set (PPS)**

A participant will be excluded from the PPS Immunogenicity analysis under the conditions presented in Table 3:

Table 3: Protocol deviations mapping and exclusion from analysis sets

| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| Informed Consent<br>Criteria | 1A - Signed informed consent/assent not available on site | All |
| | 1B - Wrong informed consent/assent version signed | All |
| | 1C - Informed consent/assent not signed and/or dated by participant (parent/Legal rep) | All |

Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\\$99638a57dafd\$76D9DDEF7D8D4E7C

B4DEE6C228977964.docx


Statistical Analysis Plan


| CTMS *<br>Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 1D – Informed consent/assent not signed and/or dated by appropriate site staff | |
| | 1E - Informed consent/assent not signed prior to any study procedure | All |
| | 1OT - Other informed consent/assent deviations | All |
| | | Manual case-by-case review |
| | 3A - Not withdrawn from study after developing withdrawal criteria | All Manual case-by-case review |
| | O. Elizibilita aritaria matarata | · |
| | 2 - Eligibility criteria not met | All |
| | 7A - Study treatment not administered per protocol | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| Eligibility and Entry Criteria | 7B - Study treatment administered while contraindication | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | | Manual case-by-case review |
| | 8A - Randomization procedure (subj assigned to wrong treatment, subj rand out of order) | All |

 $\label{lem:converter} C: \ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7CB4DEE6C228977964.docx$ Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| 2.0 | 4A - Medication, excluded by the protocol, was administered | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| Concomitant Medication Criteria | 4B - Vaccine, excluded by the protocol, was administered | By visit for Day 31 and Day 211** (based on treatment administered on Day 1 and Day 181 respectively). |
| | 8G - Biological sample specimen procedures | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| 4. Laboratory<br>Assessment Criteria | 6A - Missed assessment* *when impacting lab samples | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6D - Out of Window assessment* *when impacting lab samples | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| 5. Study Procedures<br>Criteria | 3A - Not withdrawn from study after developing withdrawal criteria | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |

Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 3B – Not discontinued from study treatment | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6A - Missed assessment | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6B – Incomplete assessment | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6C – Assessment not properly performed | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6D - Out of Window assessment | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 6OT - Other assessment or time point window | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7B – Study treatment administered while contraindication | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |

Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS *<br>Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 8C – Non study treatment supply procedures | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 8D – eDiary procedures | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 8F – Post study treatment observation not done | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 8OT - Other deviation from study procedures | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | | Manual case-by-case review |
| | 9B – Adverse event of special interest | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| 6. Serious adverse | 9C - Pregnancy | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| event criteria | 9E – SAE not reported within the expected time frame | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 9F – Failure to confirm causality assessment within the expected time frame | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |

Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 9OT – Other | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 8A - Randomization procedure (subj assigned to wrong treatment, subj rand out of order) | All |
| 7. Randomization<br>Criteria | 8B - Study blinding/unblinding procedures | By visit for Day 31 and Day 211** (based on treatment administered on Day 1 and Day 181 respectively). |
| | | Manual case-by-case review |
| 8. Visit Schedule | 5A – Missed visit/phone contact | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| Criteria | 5B – Out of window visit / contact | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| 9. Investigation Product (IP) Compliance | 7A - Study treatment not administered per protocol | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7C - Wrong study treatment or assignment administered | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |

Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 7D - Expired study treatment administered | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7E - Use of study TRT impacted by temperature excursion - not reported/approved/dispensed | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7F - Study treatment not prepared as per protocol (e.g. reconstitution) | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7G - Study treatment not available at site for administration | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7H- incorrect volume given | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | 7OT - Other deviations related to wrong study treatment/administration/dose (study treatment not available at site for administration, Commercial Vx used in place of | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | study Vx, study treatment administered while contraindication) | Manual case-by-case review |
| | 6G - Out of Window - Treatment administration | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |

 $\label{lem:converter} C: \ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7CB4DEE6C228977964.docx$ Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS *<br>Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 3A - Not withdrawn from study after developing withdrawal criteria | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| 10. Efficacy Criteria | 7B - Study treatment administered while contraindication | By visit for Day 31 and Day 211 (based on treatment administered on Day 1 and Day 181 respectively) |
| | | Manual case-by-case review |
| 11. Administrative<br>Criteria | 8E – Equipment procedures | All |
| 12. Source Document<br>Criteria | 8B – Study blinding/unblinding procedures | All |
| 13. Regulatory or Ethics Approvals Criteria | 8OT – Other deviation from study procedures | All |
| | 7OT – Other deviations related to wrong study treatment/administration/dose | All |
| 14. Other Criteria | 8E – Equipment procedures | All |
| To be discussed on a case-by-case basis | 8OT – Other deviations from study procedure | All |
| | 10A- Fraudulent data | All |

Document:

Version Number: Final 5.0 Author: PPD

Statistical Analysis Plan


| CTMS * Categories | GSK Deviations Code/ Description | Visit (timepoints) where the exclusion is applicable |
|---|---|---|
| | 10B-Any other GCP non-compliance | All Manual case-by-case review |

<sup>\*</sup> CTMS = Clinical Trial Management System. Additional details can be found in PDMP.

Note: The '4. Laboratory Assessment Criteria' includes blood draws (immunogenicity) and the '5. Study Procedures Criteria' includes the vaccination procedures.

 $\label{lem:loc-converter-lamburg} Document: C:\ProgramData\activePDF\Temp\DocConverter\API\Input\$99638a57dafd\$76D9DDEF7D8D4E7C$ 

B4DEE6C228977964.docx


<sup>\*\*</sup> All visits that follow when the exclusion occurs are also excluded.

| | | DocuSign |
|---|---|---|
| Certificate Of Completion | | |
| Envelope Id: BCEFB67708CC49FABFECE6E724<br>Subject: Please DocuSign: MENABCWY(213171<br>Project Code (Enter 0 for non-billable projects): GIQVIA ID (Login ID): PPD<br>Business Unit:<br>Global Business Operations | )_SAP_Amend4-Final_05SEP2022.docx | Status: Completed |
| Source Envelope: Document Pages: 68 Certificate Pages: 5 AutoNav: Enabled Envelopeld Stamping: Disabled Time Zone: (UTC-08:00) Pacific Time (US & Can | Signatures: 4<br>Initials: 0<br>ada) | Envelope Originator: PPD One IMS Way Plymouth Meeting, 19462 PPD |
| Record Tracking | DDD | |
| Status: Original<br>9/7/2022 4:22:08 AM | Holder: PPD | Location: DocuSign |
| Signer Events | Signature | Timestamp |
| Security Level: Email, Account Authentication (Required) | Signature<br>PPD | Timestamp Sent: 9/7/2022 4:25:09 AM Viewed: 9/7/2022 4:25:45 AM Signed: 9/7/2022 4:26:04 AM |
| PPD Security Level: Email, Account Authentication | Signature PPD With Signing Authentication via DocuSign pa With Signing Reasons (on each tab): I approve this document | Sent: 9/7/2022 4:25:09 AM<br>Viewed: 9/7/2022 4:25:45 AM<br>Signed: 9/7/2022 4:26:04 AM |

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure: PPD

| Signer Events | Signature | Timestamp |
|---|---|---|
| PPD | PPD | Sent: 9/7/2022 4:25:10 AM |
| | | Viewed: 9/15/2022 1:46:04 AM |
| Security Level: Email, Account<br>(Required) | t Authentication | Signed: 9/15/2022 1:46:27 AM |

PPD

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Flectronic Record and Signature Disclosure:

Security Level: Email, Account Authentication (Required)

Sent: 9/7/2022 4:25:10 AM Viewed: 9/7/2022 4:29:14 AM Signed: 9/7/2022 4:34:01 AM

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure: PPD

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 9/7/2022 4:25:10 AM<br>9/7/2022 4:29:14 AM<br>9/7/2022 4:34:01 AM<br>9/15/2022 1:46:27 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

# **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

# Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

# **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### How to contact IOVIA:

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

# 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

# 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

# 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

# Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

# Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.